CLINICAL TRIAL: NCT06281197
Title: Does Subspinal Le Fort I Osteotomy Affect the Nasal Airway Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Selin Celebi, PhD,DDS, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/48
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Maxillofacial Abnormalities
Keywords: Subspinal Le Fort Osteotomy; Nasal airway
MeSH Terms: conditions — Maxillofacial Abnormalities | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (Experimental): In conventional group, Le Fort I osteotomy was made using a piezosurgical saw after nasal mucosa elevation as usual Le Fort I technique.
  Interventions: Procedure: Conventional
- Subspinal Group (Active Comparator): In Subspinal group, No dissection was performed between the nasal mucosa and the ANS of the patients. Osteotomy was performed in the subspinal Le Fort I group that is described by Mommaerts . A triangular osteotomy line was created between the maxilla and the ANS with a piezosurgery.
  Interventions: Procedure: Subspinal

INTERVENTIONS:
Procedure: Conventional — Le Fort I osteotomy performed with conventional Le Fort
  Other Names: Group II
  Arms: Conventional Group
Procedure: Subspinal — Osteotomy was performed in the subspinal Le Fort I group that is described by Mommaerts
  Other Names: Group I
  Arms: Subspinal Group

SUMMARY:
After the description of Le Fort fractures, maxillary osteotomies are used to correct dentofacial deformities. The profile changes on nasolabial region resulting from a Le Fort I osteotomy, also that affects nasal airway. The Subspinal Le Fort I osteotomy (SLFIO) describe to prevent undesirable soft tissue changes. In the literature, too many articles have reported the effectiveness of SLFIO in preventing nasal deformation. However, there is no study to evaluate the nasal volume or septum deviation.

DETAILED DESCRIPTION:
The purpose of this study was objectively and subjectively to compare the effect of Subspinal Le Fort I Osteotomy and Conventional Le Fort I Osteotomy on nasal airway volume and septum deviation without additional modification such as Ans Reduction, Alar Cinch Suture, V-Y closure.

Surgical procedure; Patients were underwent general anesthesia for bimaxillary orthognathic surgery.

The mucoperiosteal flap was raised to expose the bilateral infraorbital foramina, aperture pyriformis, zygomaticomaxillary, and pterygomaxillary buttress. No dissection was performed between the nasal mucosa and the ANS of the patients in Subspinal Le Fort osteotomy group.A triangular osteotomy line was created between the maxilla and the ANS with a piezosurgery. In Conventional osteotomy group, Le Fort I osteotomy was made using a piezosurgical saw after nasal mucosa elevation. In both groups, osteotomes and pterygoid plaques, nasal septum, and lateral nasal walls were separated.

Follow up:

septum deviation and nasal. airway volume value was measured and recorded in the CBCT images taken before the surgery and at the 6th month after the surgery of each patient.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-40, ASA I, without systemic disease, without any drug allergy, and without a history of NSAID use in the week before the operation.

Exclusion Criteria:

* ASA II or higher, hepatic or renal dysfunction, neuropathic disease, long-term use of NSAIDs or opioid-derived drugs, a history of allergic reaction to drugs, pain, swelling, inflammation in the head and neck region before the operation, pregnant and breastfeeding with a history of cleft lip and palate and rhinoplasty surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Septum Deviation | up to six months
  This angle value was measured and recorded in the CBCT images taken before the surgery and at the 6th month after the surgery of each patient. If the angle in the preoperative view is smaller than the angle in the postoperative view, there is a decrease in septum deviation; If it is large, it was accepted that there was an increase in septum deviation.
Evaluation of Nasal Airway | up to six months
  CBCT scans were scanned for anatomical landmarks to adjust the volume analyzed by automatic segmentation in NemoFAB. Dens endpoint of the axis and nasion were found to be the most consistent at the anterior cranial and posterior caudal borders in the mid-sagittal plane The lateral borders were determined as the most lateral part of the nasal cavity. These markers were used to define the cubic area of interest (ROI), which includes the cranial cavity up to the maxillary base. In the sagittal tomography section, the nasal airway volume was measured in cc on the section taken from the midline.

SECONDARY OUTCOMES:
nasal obstruction scale evaluation | up to six months
  The patients filled out the form about NOSE scales in the preoperative evaluation period and the postoperative 6th month, and the sum of the score values given for each question in the questionnaire was calculated and the total scores were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Selin Çelebi, Kayseri, Meligazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guenthner TA, Sather AH, Kern EB. The effect of Le Fort I maxillary impaction on nasal airway resistance. Am J Orthod. 1984 Apr;85(4):308-15. doi: 10.1016/0002-9416(84)90188-x. PMID 6585148
- [Background] Galbiati G, Maspero C, Giannini L, Guenza GC, Zanoni F, Farronato G. Orthodontic--surgical treatment and respiratory function: rhinomanometric assessment. Minerva Stomatol. 2017 Jun;66(3):91-97. doi: 10.23736/S0026-4970.17.04045-6. Epub 2017 Apr 11. PMID 28399616
- [Background] Posnick JC, Agnihotri N. Consequences and management of nasal airway obstruction in the dentofacial deformity patient. Curr Opin Otolaryngol Head Neck Surg. 2010 Aug;18(4):323-31. doi: 10.1097/MOO.0b013e32833b9d6f. PMID 20625295
- [Background] Helal HA, Ghanem MAM, Al-Badawy AM, Abdel Haleem MM, Mousa MH. Histological and Anthropometric Changes in the Aging Nose. Aesthet Surg J. 2019 Aug 22;39(9):943-952. doi: 10.1093/asj/sjy245. PMID 30247560
- [Background] Schwarz GM, Thrash WJ, Byrd DL, Jacobs JD. Tomographic assessment of nasal septal changes following surgical-orthodontic rapid maxillary expansion. Am J Orthod. 1985 Jan;87(1):39-45. doi: 10.1016/0002-9416(85)90172-1. PMID 3881034
- [Background] Kaur S, Rai S, Kaur M. Comparison of reliability of lateral cephalogram and computed tomography for assessment of airway space. Niger J Clin Pract. 2014 Sep-Oct;17(5):629-36. doi: 10.4103/1119-3077.141431. PMID 25244276
- [Background] Goncales ES, Duarte MA, Palmieri C Jr, Zakhary GM, Ghali GE. Retrospective analysis of the effects of orthognathic surgery on the pharyngeal airway space. J Oral Maxillofac Surg. 2014 Nov;72(11):2227-40. doi: 10.1016/j.joms.2014.04.006. Epub 2014 Apr 13. PMID 24985958
- [Background] Montgomery WM, Vig PS, Staab EV, Matteson SR. Computed tomography: a three-dimensional study of the nasal airway. Am J Orthod. 1979 Oct;76(4):363-75. doi: 10.1016/0002-9416(79)90223-9. PMID 291340
- [Background] Kunkel M, Hochban W. The influence of maxillary osteotomy on nasal airway patency and geometry. Mund Kiefer Gesichtschir. 1997 Jul;1(4):194-8. doi: 10.1007/BF03043550. PMID 9384792
- [Background] Erbe M, Lehotay M, Gode U, Wigand ME, Neukam FW. Nasal airway changes after Le Fort I--impaction and advancement: anatomical and functional findings. Int J Oral Maxillofac Surg. 2001 Apr;30(2):123-9. doi: 10.1054/ijom.2000.0001. PMID 11405447
- [Background] Turvey TA, Hall DJ, Warren DW. Alterations in nasal airway resistance following superior repositioning of the maxilla. Am J Orthod. 1984 Feb;85(2):109-14. doi: 10.1016/0002-9416(84)90002-2. PMID 6594051